CLINICAL TRIAL: NCT03223714
Title: An Efficacy and Safety Trial of Intravitreal Injection of Conbercept Ophthalmic Injection in Treatment of Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Conbercept Ophthalmic Injection for Patients of Central Retinal Vein Occlusion
Acronym: CRAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KH902-CRVO-CRP-1.0
Record Dates: First submitted 2017-02-08; First posted 2017-07-21 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Macular Edema; Central Retinal Vein Occlusion
Keywords: Conbercept ophthalmic injection; ME; CRVO
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conbercept (Experimental): Conbercept
  Interventions: Drug: Conbercept Ophthalmic Injection
- Conbercept or sham (Sham Comparator): Conbercept or sham
  Interventions: Drug: Conbercept Ophthalmic Injection; Drug: sham injection

INTERVENTIONS:
Drug: Conbercept Ophthalmic Injection — Subject receive 0.5 mg Conbercept injection into their study eyes every month (Day 0 - Month 5).
  If subjects meets the criteria for repeated administration, the subject receives 0.5 mg Conbercept injection into the study eye (Month 6 ~ 11).
Drug: sham injection — Subjects receive sham injection into their study eyes every month (Day 0 - Month 5).
  Subjects receive a single intravitreal injection of 0.5 mg Conbercept ophthalmic injection in month 6, followed monthly review, if he/she meets the criteria for repeated administration, the subject receives 0.5 mg Conbercept injection into the study eye (Month 6 ~ 11).
  Arms: Conbercept or sham

SUMMARY:
This study evaluates the efficacy and safety of Conbercept ophthalmic injection. This is a multi-center, randomized, double-masked, placebo-controlled phase III clinical study. 237 patients with central retinal vein occlusion(CRVO) are expected to be enrolled in the study and randomly assigned into the Conbercept ophthalmic injection treatment group or the control group at a ratio of 2:1.

DETAILED DESCRIPTION:
The trial is divided into core and extension periods.

1. Core period (Day 0 - Month 5): Eligible subjects after the screening are assigned into the group to receive either intravitreal injection of Conbercept ophthalmic injection at a dose of 0.5 mg (treatment group) or a sham injection (control group) into their study eyes every month (Day 0 - Month 5). At month 6, primary endpoint are judged by investigators.
2. Extension period (Month 6 ~ 12): Subjects in treatment group are reviewed monthly, if he/she meets the criteria for repeated administration, the subject receives 0.5 mg Conbercept injection into the study eye (Month 6 ~ 11). Subjects in control group receive a single intravitreal injection of 0.5 mg Conbercept ophthalmic injection in month 6, followed monthly review, if he/she meets the criteria for repeated administration, the subject receives 0.5 mg Conbercept injection into the study eye (Month 6 ~ 11). The final evaluation is performed at the end of Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have signed informed consent and agreed to be followed up as per the trial protocol;
2. Aged ≥ 18 years, male or female;
3. Target eyes must meet all of following requirements:

   * Suffering from macular edema secondary to CRVO or HRVO that involves the fovea and has been first diagnosed within previous 12 months;
   * Best corrected visual acuity (BCVA) ≥24 and ≤73 letters (Snellen equivalent is 20 / 320-20 / 40);
   * Central retinal thickness (CRT) on OCT is ≥300 μm;
4. Without opacities in the refractive media and pupillary miosis that affects fundus examination.

Note: If both eyes of a subject meet the inclusion criteria, the target eye shall be determined by investigators from a medical point of view.

Exclusion Criteria:

Patients who present with any the following ocular conditions:

- Study eyes

1. Active retinal or iris neovascularization;
2. Epiretinal membrane or vitreomacular traction that investigators consider likely to affect central vision;
3. Other ocular diseases or conditions that may affect the recovery of the macula functions based on the opinion of investigators, such as foveal atrophy, foveal hemorrhage, foveal hard exudates, or dense submacular hard exudates, etc.;
4. History of retinal detachment;
5. Suffering from non-RVO diseases that may result in macular edema, visual acuity loss or retinal neovascularization during the study period based on the opinion of investigators, such as wet AMD, diabetic retinopathy, uveitis or other ocular inflammatory diseases, neovascular glaucoma, and cystoid macular edema, etc.;
6. Patients with cataract whose eye is likely to require cataract surgery within the next 12 months;
7. Have received intraocular injection of corticosteroid within previous 3 months, received subconjunctiva injection of corticosteroid within previous 6 months, or received ocular corticosteroid therapy within previous 1 month;
8. Have undergone any of the following ocular surgeries: scleral buckling surgery, PDT, vitrectomy, radial optic neurotomy or sheathotomy, glaucoma filtration surgery, parafoveal photocoagulation, pan-retinal photocoagulation, and macular translocation surgery, etc.;
9. Have received YAG laser surgery or any other ocular surgery (which including cataract surgery, macular grid photocoagulation, local retinal photocoagulation, and corneal implantation, etc.) within previous 3 months;
10. Improvement of BCVA>10 letters during screening period (comparing BCVA that is measured within 24h before first administration (Day 0) to that measured at enrollment);
11. Without lens (excluding intraocular lens) or with posterior lens capsule defect (excluding YAG laser capsulotomy following intraocular lens implantation);

    - Either eye of patients：
12. Suffering from active periophthalmitis or ocular inflammation (such as blepharitis, infectious conjunctivitis, keratitis, scleritis, uveitis and endophthalmitis, etc.);
13. Had or have uncontrollable glaucoma (defined as intraocular pressure remains ≥30 mmHg after anti-glaucoma treatment), or study eye with the cup-to-disc ratio > 0.8 due to severe glaucoma;
14. Have received anti-VEGF medications (such as Lucentis, Avastin, or Conbercept, etc.) within 3 months before screening;

    - Patients who present with any the following systematic conditions:
15. Patients have allergic reaction or history of allergy to sodium fluorescein, have a history of allergy to protein products for therapy or diagnosis, and are sensitized to two or more drugs and/or non-drug factors, or suffering from allergic diseases;
16. Patients with a history of stroke, or with a history of myocardial infarction and/or cerebrovascular disease or a history of transient cerebral ischemia within 6 months before screening, or with active disseminated intravascular coagulation and significant bleeding tendencies;
17. Patients who are diagnosed with systemic autoimmune diseases (such as ankylosing spondylitis, systemic lupus erythematosus, Behcet's disease, rheumatoid arthritis, and scleroderma, etc.)；
18. Patients who are diagnosed with any clinically uncontrollable disease (such as HIV, active hepatitis, metabolic disorders, severe mental, neurological, cardiovascular, respiratory and other diseases and cancer);
19. Hypertensive patients whose blood pressure have not been controlled effectively (defined as SBP ≥160 mmHg or DBP ≥100 mmHg after treatment with antihypertensive drugs);
20. Patient who has a surgical history within 1 month before enrollment, and/or is currently suffering from unhealed wounds, ulcers, fractures, etc.;
21. Use of systemic (orally, intramuscularly or intravenously) corticosteroids within 6 months before screening;
22. Patients received systemic anti-VEGF medications (such as Avastin) within 6 months before screening; Patients underwent laboratory test with any of the following abnormal results
23. Liver, kidney and immune dysfunction (defined as ALT and AST ≥ 2 × UNL of the laboratory , Crea and BUN ≥ 1.5 × UNL of the laboratory in the site of this trial);
24. Coagulation abnormalities (prothrombin time ≥ 3 seconds + UNL, and active partly thromboplastin time ≥ 10 seconds + UNL);

    Patients of childbearing age under any of the following conditions:
25. Do not use an effective method of contraception;

    Note: subject with the following conditions are not excluded:
    * 12 months of amenorrhea for natural reasons, or 6 months of natural amenorrhea for natural reasons and levels of serum follicle stimulating hormone <40mlU/ml;
    * 6 weeks after ovariectomy of both sides with / without concurrent hysterectomy;
    * Use one or more acceptable birth control methods as follows:

    Sterilization (male companion has undergone bilateral vasectomy or resection) Hormonal birth control (implantable, patch or oral route) Intrauterine device and double barrier methods
    * Take reliable birth control measures throughout the study period, and continuously do so for 30 d after stopping study medication (unacceptable birth control methods including periodic abstinence, calendar-based method, ovulation phase method, body temperature measurement, luteal phase method and onanism);
26. Pregnant and breast-feeding women. Pregnancy is defined as a positive urine pregnancy test in this trial; Others
27. Participate in any drug (exclusive of vitamins and minerals) clinical trial within 3 months prior to the screening (if the investigational drug has a long half-life, 3 months or 5 half-lives, whichever is longer);
28. The Subject is otherwise determined by the Investigator to be medically unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | month 6
  To compare mean changes in Best Corrected Visual Acuity (BCVA) from baseline between the Conbercept ophthalmic injection treatment group (treatment group) and the control group at month 6.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | month 3 and month 12
  To evaluate mean changes in BCVA from baseline of the treatment group and the control group at month 3 and 12.
Central Retinal Thickness | month 3, month6 and month 12
  To evaluate mean changes in Central Retinal Thickness (CRT) from baseline of the treatment group and the control group at month 3, 6 and 12.
Number of subject who received laser rescue treatment | month 6 and month 12
  To evaluate the number of subjects who received laser rescue treatment of the treatment group and the control group at month 6 and 12.
Number of participants with treatment-related the systemic and ocular safely as assessed | month 6 and month 12 or trail period
  To evaluate the systemic and ocular safety of the treatment group and the control group.

OTHER OUTCOMES:
distribution of BCVA changes | month 3, month 6 and month 12
  To evaluate the distribution of BCVA changes from baseline of the treatment group and the control group at month 3, 6 and 12.
Mean change in Best Corrected Visual Acuity | month 0,month 1,month 2,month 3,month 4,month 5,month 6,month 7,month 8,month 9,month 10,month 11 and month 12
  To evaluate mean changes in BCVA from baseline of the treatment group and the control group at every visit for 1 year.
Mean changes in CRT, Macular Volume | month 0,month 1,month 2,month 3,month 4,month 5,month 6,month 7,month 8,month 9,month 10,month 11 and month 12
  To evaluate the average changes in imaging findings (e.g., CRT and total macular volume) relative to the baseline for treatment group and control group at each follow-up visit for 1 year

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Beijing Friendship Hospital,Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The General Hospital of the People's Liberation Army, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Army Medical Center, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - Zhongshan Ophthalmic Center, Guangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - The Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing First Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Eye & Ent Hospital of Fudan University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital School of Optometry & Eye Institute, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Eye Hospital,WMU Zhejiang Eye Hospital, Wenzhou
  - Wuhan General Hospital of Guangzhou Military Command, Wuhan
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an